CLINICAL TRIAL: NCT03238443
Title: Interest of the Donor-specific and Complement-binding Anti-HLA Antibodies (C1q) Assays for the Management and the Monitoring After Liver Transplant
Brief Title: Interest of the Donor-specific Antibodies After Liver Transplantation
Acronym: vaLIDLIver
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2014_18; 2015-A00418-41 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-07-31; First posted 2017-08-03 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Liver Transplant
Keywords: DSA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a prospective observational mono center study

Primary objective :

Study the anti-HLA antibodies frequency preformed before liver transplantation and the kinetic of appearance of DSA and de novo complement-binding anti-HLA antibodies after liver transplantation.

Secondary objective :

* Risk factor of de novo DSA appearance (Immunosuppressive therapy, liver aetiology)
* Impact of DSA on:

  * Graft and patients survivals
  * Onset of allograft rejection (acute, late-onset, chronic)
  * Unexplained liver graft dysfunction
  * Unexplained liver enzymes abnormalities
  * Liver fibrosis development (liver stiffness study using fibroscan©)

ELIGIBILITY:
Inclusion Criteria:

* Liver transplanted patients older than 18, transplanted in Lille University Hospital.
* Written consent by the patient or his/her legal representative (especially patient with hepatic encephalopathy).
* Patients with health insurance

Exclusion Criteria:

* Minor patients.
* Pregnant women or during lactation.
* Patient under curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients transplanted at the University Hospital of Lille will be included in a prospective observational study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2019-07-13 (Actual); Study Completion 2019-07-13 (Actual)

PRIMARY OUTCOMES:
Prevalence DSA positivity (or anti-HLA). | At baseline
  The positivity is defined as a fluorescence ≥ 1000.

SECONDARY OUTCOMES:
Fluorescence quantification | at 3 months, 1 year and 2 years after transplantation
Presence of C1q binding-complement anti-HLA antibodies | at 3 months, 1 year and 2 years after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Dharancy, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU, Hôpital Claude Huriez, Lille, France

IPD SHARING:
Plan to Share IPD: No